CLINICAL TRIAL: NCT02848287
Title: Influence of 0.75% Ropivacaine Topicalization on Emergence Agitation in Preschool-aged Children Undergoing Adenotonsillectomy
Brief Title: Influence of 0.75% Ropivacaine Topicalization on Emergence Agitation in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Go Un Roh, Clinical assistant professor, primary investigator, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-DRU-16-061
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Saline Solution; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): 1*2 gauze is soaked with 5 cc of 0.9 % normal saline, applied in tonsillar fossae for 3 min, then removed.
  Interventions: Drug: normal saline
- Ropivacaine (Experimental): 1*2 gauze is soaked with 5 cc of 0.75% ropivacaine, applied in tonsillar fossae for 3 min, then removed.
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: normal saline — 1*2 gauze is soaked with 5 cc of 0.9 % normal saline, applied in tonsillar fossae for 3 min, then removed.
  Arms: Normal Saline
Drug: ropivacaine — 1*2 gauze is soaked with 5 cc of 0.75% ropivacaine, applied in tonsillar fossae for 3 min, then removed.
  Arms: Ropivacaine

SUMMARY:
Emergence agitation (EA) is highly prevalent in children after surgery. Risk factors for EA are Eye, nose and throat (ENT) surgery, preoperative anxiety, postoperative pain. There are several preventive strategies but none of them completely prevent EA.

Topical application of ropivacaine can reduce post-tonsillectomy pain. Therefore, it might reduce the incidence of postoperative EA.

ELIGIBILITY:
Inclusion Criteria:

* American Society of anesthesiologist physical status class I/II
* tonsillectomy or adenotonsillectomy under general anesthesia

Exclusion Criteria:

* obstructive sleep apnea
* developmental delay attention deficit hyperactivity disorder, allergy to local anesthetics, convulsion disorder

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Paediatric anesthesia emergence delirium scale (PAED) score at PACU admission | 1 min after postanesthesia care unit (PACU) admission
  PAED score is assessed

SECONDARY OUTCOMES:
Face legs activity cry consolability (FLACC) score | 1 min after postanesthesia care unit (PACU) admission
  FLACC score is assessed.
PAED score 10 min after PACU admission | 10 min after postanesthesia care unit (PACU) admission
PAED score 20 min after PACU admission | 20 min after postanesthesia care unit (PACU) admission
PAED score 30 min after PACU admission | 30 min after postanesthesia care unit (PACU) admission
FLACC score 10 min after PACU admission | 10 min after postanesthesia care unit (PACU) admission
FLACC score 20 min after PACU admission | 20 min after postanesthesia care unit (PACU) admission
FLACC score 30 min after PACU admission | 30 min after postanesthesia care unit (PACU) admission

IPD SHARING:
Plan to Share IPD: No